CLINICAL TRIAL: NCT04088786
Title: Phase I Trial of Cytoreductive Surgery and Heated Intraperitoneal Chemotherapy With Nanoliposomal Irinotecan in Patients With Peritoneal Surface Malignancies
Brief Title: Phase I Trial HIPEC With Nal-irinotecan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Ipsen (Industry); Barbara Ann Karmanos Cancer Institute (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, minsig Choi, Clinical Associate Professor of Medicine, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00059 HIPEC Nal-IRI
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Peritoneal Cancer; Pseudomyxoma Peritonei; Mucinous Adenocarcinoma; Mucinous Tumor; Colorectal Cancer; Gastric Cancer; Primary Peritoneal Carcinoma; Mesothelioma
Keywords: HIPEC; nal-irinotecan
MeSH Terms: conditions — Pseudomyxoma Peritonei; Adenocarcinoma, Mucinous; Neoplasms, Cystic, Mucinous, and Serous; Colorectal Neoplasms; Stomach Neoplasms; Mesothelioma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Intervention Model Description: This is a 3+3 dose-finding cohort design.
Masking Description: All eligible patients will be treated with the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Experimental): Cytoreductive surgery (CRS) followed by study treatment with nanoliposomal irinotecan administered intraperitoneally.
  Interventions: Drug: nanoliposomal irinotecan

INTERVENTIONS:
Drug: nanoliposomal irinotecan — The starting dose of nal-IRI will be 70 mg/m2 (cohort level 1) applied for 30 min using a closed HIPEC technique following completion of cytoreductive surgery. If there is dose limiting toxicity (DLT) in cohort level 1, then the dose will be reduced the dosage of the next cohort to 50 mg/m2 (cohort level 0). If there is no DLT, the dose of nal-IRI will be increased to 140 mg/m2, 210 mg/m2 and 280 mg/m2 . If one of the patients experiences DLT, then the cohort will expand to 6 patients and accrual to the current dose level and dose escalation will stop if 2 or more patients experience a DLT at a given dose level.

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of intraperitoneal administration of heated nanoliposomal Irinotecan in cytoreductive surgery (CRS), which is surgery designed to remove as much of the cancer as possible, and heated intraperitoneal chemotherapy (HIPEC) procedures.

DETAILED DESCRIPTION:
Cytoreductive surgery and heated intraperitoneal chemotherapy consists of two parts: the first is the surgical removal of all grossly visible deposits of cancer from the abdomen; and the second is application of heated chemotherapy in salt water at the same time as the removal of the visible cancer. HIPEC is an alternative method of delivering chemotherapy. Traditional chemotherapy is injected into a vein, while HIPEC applies chemotherapy drugs warmed up by an FDA-approved machine to 108 degrees Fahrenheit directly into the abdomen during surgery, making it an option for cancers that originated in or have spread to the abdominal cavity. Standard treatment in this manner usually includes Mitomycin C or Cisplatin as its chemotherapy agents. In this study, the investigators will use nanoliposomal irinotecan as the chemotherapy agent. Irinotecan is FDA approved for the treatment of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pseudomyxoma peritonei or peritoneal carcinomatosis of digestive origin or primary peritoneum: appendiceal mucinous tumor or adenocarcinoma (including goblet cell cancer and signet ring cell cancer), colorectal cancer, gastric cancer, primary peritoneal adenocarcinoma, and mesothelioma; regardless of the number of prior treatment lines. Diagnosis of peritoneal metastasis to be confirmed via either clinical or histopathology assessment.
2. Age ≥18 years
3. Eastern Cooperative Oncology Group performance status of 0 or 1
4. Patients must be candidates for grossly complete cytoreduction surgery with life expectancy greater than 3 months
5. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count >1,500/microliter (mcL) and white blood cells > 4000/mm3
   * platelets >75,000/microliters
   * total bilirubin < 3x upper limit normal for institutional limits
   * aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) <2.5x institutional upper limit of normal
   * creatinine within normal institutional limits
6. Documentation of resectable disease extent by radiographic peritoneal carcinomatosis index (PCI) score or preoperative diagnostic surgery/laparoscopy with preoperative measurements taken within 6 weeks of study entry.
7. Women of child-bearing potential and men must agree to use adequate contraception (barrier or hormonal plus barrier method of birth control; abstinence) prior to study entry and for the duration of study participation (at least first 6 months). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with peritoneal disease considered to be unresectable according to preoperative clinical criteria.
2. Patients who undergo debulking for palliation with persistence of gross residual disease (complete of cytoreduction score 3, CC=3) will be ineligible for the study.
3. Large burden visceral metastases or extra-abdominal metastases.
4. Patients who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. There is no limit on the number of prior lines of chemotherapy.
5. Patients may not be receiving any other investigational agents.
6. History of allergic reactions to nal-IRI or irinotecan.

7 Uncontrolled ongoing illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

8 Pregnant or breast-feeding women are excluded from this study.

9 HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 4 weeks post surgery
  To assess the safety and feasibility of administering nanoliposmal irinotecan intraperitoneally following cytoreductive surgery.

SECONDARY OUTCOMES:
Plasmatic dosages | 48 hours
  Determine the correlation of intraperitoneal dosages of nanoliposomal irinotecan with plasma blood levels using pharmacokinetic analysis
Disease Free survival | 6 months
  Assess the efficacy of intraperitoneal administration of nanoliposomal irinotecan relating to disease free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Minsig Choi, MD, Principal Investigator — Stony Brook University; Joseph Kim, MD, Principal Investigator — University of Kentucky; Georgios Georgakis, MD, Principal Investigator — Stony Brook University
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Stony Brook University Cancer Center, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald HG, Cassim EB, Harper MM, Burke EE, Marcinkowski EF, Cavnar MJ, Pandalai PK, Kim J. The Development of Investigator-Initiated Clinical Trials in Surgical Oncology. Surg Oncol Clin N Am. 2023 Jan;32(1):13-25. doi: 10.1016/j.soc.2022.07.003. Epub 2022 Nov 3. PMID 36410913